CLINICAL TRIAL: NCT00391222
Title: A Randomized, Double Blind, Placebo and Active Controlled Parallel Group Study to Evaluate the Efficacy and Safety of Risperidone Long-acting Injectable (LAI) for the Prevention of Mood Episodes in the Treatment of Subjects With Bipolar I Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Risperidone for the Prevention of Mood Episodes in the Treatment of Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR012145; NCT01205113 (obsolete NCT alias)
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder; Intramuscular injection; prevention of mood episodes; long acting injectable; risperidone
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): Risperidone Long Acting Injectable (LAI) Intramuscular injections of risperidone LAI (25 37.5 or 50 mg) every 2 weeks and oral placebo daily
  Interventions: Drug: Risperidone Long Acting Injectable (LAI)
- 002 (Placebo Comparator): Placebo Intramuscular injections of placebo every 2 weeks and oral placebo daily
  Interventions: Drug: Placebo
- 003 (Active Comparator): Olanzapine Intramuscular injections of placebo every 2 weeks and oral olanzapine 10 mg daily
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Intramuscular injections of placebo every 2 weeks and oral olanzapine 10 mg daily
  Arms: 003
Drug: Placebo — Intramuscular injections of placebo every 2 weeks and oral placebo daily
  Arms: 002
Drug: Risperidone Long Acting Injectable (LAI) — Intramuscular injections of risperidone LAI (25, 37.5, or 50 mg) every 2 weeks and oral placebo daily
  Arms: 001

SUMMARY:
The purpose of this randomized, double blind, double dummy, multicenter study was to evaluate the efficacy of risperidone long-acting injectable (LAI) monotherapy in comparison with placebo in the prevention of a mood episode in treatment of patients with bipolar I disorder. Oral olanzapine was used to assess the validity of the study design. The primary objective of this study is to evaluate the efficacy of risperidone LAI versus placebo in the prevention of a mood episode (recurrence event) in patients with bipolar I disorder after a 12-week (3 month) stabilization period on risperidone LAI, as measured by the time to recurrence of any mood episode. Risperidone LAI has been approved by the FDA in the USA for the treatment of patients with schizophrenia and for the prevention of mood recurrences in bipolar I disorder, as monotherapy or add-on treatment. It is approved at EMEA and other European and non-European health authorities for the treatment of patients with schizophrenia, too.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy multicenter study with 3 parallel arms (risperidone long-acting injectable (LAI), placebo, and olanzapine) to evaluate the efficacy and safety of risperidone LAI versus placebo in the prevention of a mood episode (recurrence event). The primary objective of this study is to evaluate the efficacy of risperidone LAI monotherapy versus placebo in the prevention of a mood episode (recurrence event) in patients with bipolar I disorder after a 12-week (3 month) stabilization period on risperidone LAI, as measured by the time to recurrence of any mood episode. This study includes 3 periods - the screening period (Period I, lasting up to 2 weeks); the open-label treatment period (Period II, lasting 12 weeks); and the double-blind treatment period (Period III, lasting up to 18 months and at least 9 months). In the open -label treatment period (Period II) treatment with risperidone LAI will be started with injection of a recommended dose of 25 mg every 14 days in patients entering Period II. If judged clinically appropriate, patients may start with 37.5 mg every 14 days. Dosage can only be increased (up to a maximum dose of 50 mg every 14 days) if the Clinical Global Impression - Severity (CGI-S) score has increased by => 1 over 2 consecutive assessments at least 2 weeks apart and if there is symptom exacerbation that cannot be treated adequately with short-term (14 days) benzodiazepine medication. If an increase in risperidone LAI dosage is necessary, oral risperidone (1 to 2 mg/day) needs to be added for 3 weeks after the first injection of the higher dosage. Washout of all psychotropics other than risperidone long acting must be completed by the end of the first week. Non-acute patients on an antipsychotic or mood stabilizer for at least 4 weeks will continue their previous treatment for the first 3 weeks. No changes will be made in the regimens of non-acute patients receiving an antipsychotic or mood stabilizer unless there is concern about efficacy or safety.Patients experiencing an acute manic or mixed episode will additionally be treated with oral risperidone at whole-milligram dosages between 1 and 6 mg/day as needed to treat the symptoms of the acute episode for the first 3 weeks, in order to cover the 3 weeks lag period of Risperidone long acting. Patients experiencing an acute episode who do not respond to treatment within 4 weeks will be discontinued from the study. Patients who do not show a response (acute patients at baseline) or do not maintain the efficacy (non-acute patients at baseline and acute patients after initial response) during the 12-week (3 month) open-label risperidone LAI stabilization period (Period II), will be discontinued from the study as soon as any one of the following criteria is met: The patient meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, text revised (DSM-IV-TR) criteria for a hypomanic, manic, mixed, or depressive episode; the patient needs treatment intervention with any mood stabilizer, antipsychotic medication (other than study drug), benzodiazepine (beyond the dosage allowed), or antidepressant medication; the patient requires hospitalization for any bipolar mood episode; the patient either has a Young Mania Rating Scale (YMRS) score >12 in combination with CGI-S score =>4 or a Montgomery-Åsberg Depression Rating Scale (MADRS) score >12 in combination with a CGI-S score =>4. (If either of these criteria is fulfilled at an assessment but if the investigator assumes that this is only a temporary state that requires no action, the investigator is allowed to postpone the decision about maintenance or response by a maximum of 4 days. If after 4 days, the criteria are still met, the patient must be withdrawn from Period II.) Patients who show initial and maintained response (acute patients at baseline) or who maintain the efficacy (non-acute patients at baseline) during the 12-week (3-month) open-label risperidone LAI stabilization period (Period II), will be eligible for entering the double-blind treatment period (Period III). Patients who enter Period III will be randomized to receive intramuscular injections of risperidone LAI every 14 days (at the dosage achieved at the end of Period II) and oral placebo daily, or placebo injections every 14 days and oral placebo daily, or placebo injections every 14 days and oral olanzapine 10 mg/day. No supplementation with oral risperidone and no dosage titration will be allowed during this period of the study. Using the double-dummy design, all patients will receive an intramuscular injection every 14 days and will take oral medication every day. Patients who present with a recurrence during Period III, will be considered as meeting the end point of the study. Patients will remain in the double-blind treatment period until they meet recurrence criteria, until they withdraw consent, or are lost to follow-up, until the last patient completed at least 9 months without a mood episode in Period III, or until the study ends. The study will end when 158 patients have presented with a mood episode in Period III, or if the study is terminated based on the decision of the sponsor. Approximately 860 patients meeting the inclusion and exclusion criteria will be enrolled in this study, with the goal of observing at least 158 recurrence events in Period III. Safety evaluations will include adverse events, clinical laboratory tests - including blood glucose/lipid profile (fasting), prolactin, TSH, and urinalysis - vital signs (pulse and blood pressure) and ECG, physical examination, body weight and height, the Extrapyramidal Symptom Rating Scale, pregnancy testing, and urine drug screen. The patients will receive risperidone LAI (25, 37.5 or 50 mg (period II)) every 14 days during the 12 week long open-label period (Period II). Patients who enter the double-blind period (Period III) will be randomized to receive intramuscular injections of risperidone LAI every 14 days and oral placebo daily, or placebo injections every 14 days and oral placebo daily, or placebo injections every 14 days and oral olanzapine 10 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I disorder as defined by DSM-IV-TR criteria. All diagnoses will be confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I.). Patients who present with additional signs or symptoms compatible with Axis I diagnoses of social anxiety disorder or generalized anxiety disorder are acceptable. All other comorbid or active Axis I diagnoses are excluded. Personality disorders as defined by DSM IV TR criteria are acceptable, with the exception of antisocial and borderline personality disorders
* Must be currently experiencing a manic or mixed episode (acute
* YMRS >20 and CGI-S =>4 [moderate]) or must be between mood episodes (non-acute
* YMRS <12 and CGI-S=<3 [mild])
* Must have had at least 2 bipolar mood (manic, mixed manic, or depressed) episodes, exclusive of the current episode (if applicable), during the last year. For non-acute subjects (YMRS <12 and CGI-S=<3 [mild]), one manic episode must have occurred within 4 months of enrollment
* Patients who are non-acute (YMRS <12 and CGI-S =<3 [mild]) and are currently receiving an antipsychotic other than risperidone or a mood stabilizer must have received this other medication at the same dosage for a minimum of 4 weeks and must be either experiencing problems of safety or tolerability with the antipsychotic or mood stabilizer or request a change of medication

Exclusion Criteria:

* No history of more than 4 mood episodes each year (rapid cycling) during the last 2 years prior to screening
* No history of ADHD, anxiety disorder, or panic disorder as the primary diagnosis
* Not meeting DSM-IV-TR criteria for a hypomanic or depressive episode
* Not meeting DSM-IV-TR criteria for any comorbid or active Axis I disorder other than those specifically allowed in the Inclusion Criteria
* Not meeting DSM-IV-TR criteria for antisocial or borderline personality disorder
* Not having a chronic or serious general medical illness, including hepatic, renal, respiratory, cardiovascular, endocrine, neurologic (including seizure disorder), or hematologic disease as determined by the clinical judgment of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (63):
- China (7):
  - Baoding
  - Beijing
  - Guangzhou
  - Nanjing
  - Shanghai
  - Suozhou
  - Wuhan
- Colombia (6):
  - Barranquilla Atlantico
  - Bello Antioquia
  - Bogotá
  - Bogotá S/N
  - Medellin Antioquia
  - Pereira Risaralda
- Germany (3):
  - Freiburg im Breisgau
  - Hildesheim
  - Oranienburg
- Athens, Greece
- India (10):
  - Ahmedabad
  - Bangalore
  - Chennai
  - Hyderabad
  - Ludhiana
  - Mangalore
  - Mumbai
  - New Delhi
  - Pune
  - Varanasi
- Jakarta, Indonesia
- Amman, Jordan
- Beirut, Lebanon
- Malaysia (2):
  - Johor Bahru
  - Kuala Lumpur
- Mexico (7):
  - Mexico City
  - Mérida
  - Monterrey
  - Puebla City
  - Tabasco
  - Tampico
  - Zapopan
- Peru (2):
  - Lima
  - Lima Lima
- Philippines (3):
  - Iloilo City
  - Mandaluyong
  - Mandaue City
- Russia (13):
  - Arkhangelsky District
  - Chelyabinsk
  - Izhevsk
  - Kazan’
  - Moscow
  - Moscow Region
  - Nizny Novgorod
  - Orenburg
  - Saint Petersburg
  - Saratov
  - Stavropol Na
  - Tomsk Na
  - Voronezh
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Durban
  - Pretoria
- Taiwan (2):
  - Tainan
  - Taipei

REFERENCES:
- See also: A randomized, double-blind, placebo and active-controlled, parallel-group study to evaluate the efficacy and safety of risperidone long-acting injectable for the prevention of mood episodes in the treatment of subjects with bipolar I disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=26&filename=CR012145_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was run from 14 November 2006 to 13 April 2009. Patients were recruited at 70 investigational sites located in 14 countries across Europe, Asia, Latin-America, and Africa.
Pre-assignment Details: Patients were treated appropriately or continued previous treatment. At baseline, treatment with Risperidone Long Acting Injectable (LAI) was started. During 12 weeks patients were stabilized on risperidone LAI and treatment with antipsychotics, mood stabilizers and other psychotropics was titrated off unless otherwise specified in the protocol.
Groups:
- Risperidone LAI: Double-blind Period III: risperidone long-acting injectable 25, 37.5 or 50 mg intramuscular every 14 days and oral placebo daily
- Placebo: Double-blind Period III: placebo injections every 14 days and oral placebo daily
- Olanzapine: Double-blind Period III: placebo injections every 14 days and oral olanzapine daily
- Open-label Risperidone LAI: Open-label Period II: risperidone long-acting injectable 25, 37.5 or 50 mg intramuscular every 14 days
Period: Period II (Open-label Risperidone LAI)
Arm/Group | Risperidone LAI | Placebo | Olanzapine | Open-label Risperidone LAI
Started | 0 | 0 | 0 | 560 (The 25 patients at the site of Dr. Parikh were excluded from the analysis due to GCP non-compliance)
Completed | 0 | 0 | 0 | 398
Not Completed | 0 | 0 | 0 | 162
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 26
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 10
Not completed — Non-responder | 0 | 0 | 0 | 97
Not completed — Other | 0 | 0 | 0 | 24
Period: Period III (Double-Blind Treatment)
Arm/Group | Risperidone LAI | Placebo | Olanzapine | Open-label Risperidone LAI
Started | 132 (Patients were randomized to one of 3 arms in Period III, after completing open-label Period II) | 135 (Patients were randomized to one of 3 arms in Period III, after completing open-label Period II) | 131 (Patients were randomized to one of 3 arms in Period III, after completing open-label Period II) | 0
Completed | 104 | 113 | 108 | 0
Not Completed | 28 | 22 | 23 | 0
Not completed — Withdrawal by Subject | 15 | 12 | 6 | 0
Not completed — Lost to Follow-up | 2 | 4 | 4 | 0
Not completed — Adverse Event | 5 | 2 | 4 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 0
Not completed — Study Medication Non-compliant | 0 | 1 | 3 | 0
Not completed — Other | 6 | 1 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risperidone LAI: Double-blind Period III: risperidone long-acting injectable intramuscular every 14 days and oral placebo daily
- Olanzapine: Double-blind Period III: placebo injections every 14 days and oral olanzapine 10 mg/day
- Total: Total of all reporting groups
Arm/Group | Risperidone LAI | Placebo | Olanzapine | Total
Number analyzed (Participants) | 132 | 135 | 131 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.76 (11.23) | 36.87 (11.08) | 36.57 (11.10) | 36.41 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 71 | 59 | 208
  Male | 54 | 64 | 72 | 190

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence of a Mood Episode (Risperidone LAI Versus Placebo)
Description: Recurrence was estimated using the Kaplan-Meier method and defined as meeting any of the following: DSM-IV-TR criteria for a hypomanic, manic, mixed, or depressive episode; in need of mood stabilizer, antipsychotic medication, benzodiazepine or antidepressant; requiring hospitalization for mood episode; either Young Mania Rating Scale (YMRS) >12 or Montgomery-Åsberg Depression Rating Scale (MADRS) >12 combined with Clinical Global Impression - Severity (CGI-S) >=4; in need of increase in study medication dose or supplementation with oral risperidone or another antipsychotic or mood stabilizer.
Time Frame: Assessed at every visit from the moment of randomization to a treatment arm (baseline Period III) until the end of treatment (Month 21 or earlier)
Population: ITT analysis set for Period III: all randomized patients who received at least one dose of double-blind study medication and who had at least one post-baseline visit. This excluded 2 patients in both the risperidone LAI arm (discontinued the study due to withdrawal of consent or adverse event) and placebo arm (both withdrew consent).
Measure: Mean (Standard Error); unit: days
Arm/Group | Risperidone LAI | Placebo
Number analyzed (Participants) | 131 | 133
days | 293.39 (15.93) | 270.47 (17.74) [171 to 354]
Statistical Analysis 1: Comparison: Risperidone LAI vs Placebo; Comparison between risperidone LAI and placebo was performed using a log-rank test controlling for patient type at screening (acute or non-acute) and for geographic region. As recurrence rates at 9 months were assumed to be 45% for risperidone LAI and 68% for placebo, the study would have approximately 90% power to detect a clinically meaningful difference of 23% in recurrence rates of a mood episode if in Period III 100 patients were randomized to each of the 2 relevant treatment arms; Test type: Superiority or Other; p = 0.057, Log Rank — As defined in the protocol, the olanzapine arm was not included in the primary outcome comparison. Data on the olanzapine arm are presented in outcome measure 7

2. Secondary Outcome: Time to Recurrence of an Elevated Mood (Hypomanic, Manic, or Mixed) Episode
Description: Recurrences were classified as elevated mood or depressive by the investigator based on the patient's data at the time of the event. Time to recurrence of an elevated mood episode was estimated by means of the same survival analysis method as for the primary outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Risperidone LAI | Placebo | Olanzapine
Number analyzed (Participants) | 131 | 133 | 130
days | 357.41 (13.94) | 323.14 (18.57) | 448.03 (12.42)
Statistical Analysis 1: Comparison: Risperidone LAI vs Placebo; The time-to-event data were evaluated by the same survival analysis method as used for the primary outcome. The recurrence rates (Kaplan-Meier estimated) were calculated for each treatment arm using the same methods as for the primary outcome; Test type: Superiority or Other; p = 0.005, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Olanzapine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Secondary Outcome: Time to Recurrence of a Depressive Episode
Description: Recurrences were classified as elevated mood or depressive by the investigator based on the patient's data at the time of the event. Time to recurrence of a depressive episode was estimated by means of the same survival analysis method as for the primary outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Risperidone LAI | Placebo | Olanzapine
Number analyzed (Participants) | 131 | 133 | 130
days | 213.86 (7.23) | 300.20 (10.64) | 356.11 (7.63)
Statistical Analysis 1: Comparison: Risperidone LAI vs Placebo; The time-to-event data were evaluated by means of the same survival analysis method as used for the primary outcome. The recurrence rates (Kaplan-Meier estimated) were calculated for each treatment arm using the same methods as for the primary outcome; Test type: Superiority or Other; p = 0.655, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Olanzapine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.011, Log Rank

4. Secondary Outcome: Time to Early Study Discontinuation for Any Reason
Description: The robustness of the primary outcome analysis was tested by means of a sensitivity analysis: patients who discontinued the study during Period III for any reason were analyzed as having a recurrence of a mood episode at the time of their study discontinuation. The same survival analysis method as for the primary outcome was applied.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Risperidone LAI | Placebo | Olanzapine
Number analyzed (Participants) | 131 | 133 | 130
days | 252.45 (15.87) | 236.14 (16.02) | 365.64 (16.16)
Statistical Analysis 1: Comparison: Risperidone LAI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2882, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Olanzapine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank

5. Secondary Outcome: Change From Double-blind Baseline to Endpoint in Young Mania Rating Scale (YMRS)
Description: The 11-item YMRS was administered by an adequately trained clinician who did not provide psychotherapy or psycho-education to the patient. A severity rating was assigned to each of the items, based on the patient's subjective report of his or her condition over the previous 7 days or since the last visit (whichever was shorter) and the clinician's behavioral observations during the interview, with emphasis on the latter. The total YMRS score included the score of all 11 items ranging from 0 to 60, a higher score indicating a more severe condition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone LAI | Placebo | Olanzapine
Number analyzed (Participants) | 131 | 133 | 130
units on a scale | 2.9 (0.86) | 8.0 (1.16) | 1.7 (0.77)
Statistical Analysis 1: Comparison: Risperidone LAI vs Placebo; An ANCOVA model was applied to the change from baseline of Period III at each time point in Period III, with treatment, patient type at screening, and geographic region as factors and baseline YMRS total score as covariate. The comparison between active treatment and placebo was performed based on the LS means obtained from the ANCOVA model. The difference in LS means between treatment arms was estimated, as was the 95% confidence interval for the difference; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Olanzapine; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Change From Double-blind Baseline to Endpoint in Montgomery Åsberg Depression Rating Scale (MADRS)
Description: The MADRS was assessed by an adequately trained clinician who did not provide psychotherapy or psycho-education to the patient. The scale consists of 10 items that cover all of the core depressive symptoms. Each item is scored from 0 to 6 and a total score is calculated by adding the scores of all 10 items. For each individual item as well as for the total score, a higher score represents a more severe condition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone LAI | Placebo | Olanzapine
Number analyzed (Participants) | 131 | 133 | 130
units on a scale | 5.1 (0.87) | 6.1 (0.99) | 2.0 (0.65)
Statistical Analysis 1: Comparison: Risperidone LAI vs Placebo; An ANCOVA model was applied to the change from baseline of Period III at each time point in Period III, with treatment, patient type at screening, and geographic region as factors and baseline MADRS total score as covariate. The comparison between active treatment and placebo was performed based on the LS means obtained from the ANCOVA model. The difference in LS means between treatment arms was estimated, as was the 95% confidence interval for the difference; Test type: Superiority or Other; p = 0.480, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Olanzapine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA

7. Secondary Outcome: Time to Recurrence of a Mood Episode (Exploratory/Olanzapine)
Description: Recurrence was defined as for the risperidone LAI and placebo arms (meeting any of 5 criteria). Since the study was designed to compare the efficacy of risperidone LAI versus placebo, this olanzapine analysis was exploratory in nature.
Time Frame: as for outcome 1
Population: ITT analysis set for Period III: all randomized patients who received at least one dose of double-blind study medication and who had at least one post-baseline visit. This excluded 1 patient in the olanzapine arm (discontinued the study due to non-compliance to the study medication).
Measure: Mean (Standard Error); unit: days
Arm/Group | Olanzapine
Number analyzed (Participants) | 130
days | 414.04 (14.78)

ADVERSE EVENTS:
Time Frame: AEs were collected from the signing of the informed consent onwards until the last study-related procedure up to 21 months or early discontinuation.
Description: The AEs described hereafter are treatment-emergent AEs, defined as having their onset in the specific treatment period in which they were reported and up to 45 days after the last dose of study medication, given the long half-life of risperidone LAI.
Groups:
- Risperidone LAI: Double-blind Period III: risperidone LAI 25, 37.5 or 50 mg intramuscular every 14 days and oral placebo daily
- Open-label Risperidone LAI: risperidone 25, 37.5, or 50 mg intramuscular every 14 days
Arm/Group | Risperidone LAI | Placebo | Olanzapine | Open-label Risperidone LAI
Serious Adverse Events (participants affected / at risk) | 19/132 | 32/135 | 13/131 | 34/560
Other Adverse Events (participants affected / at risk) | 90/132 | 77/135 | 96/131 | 326/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone LAI (N=132) | Placebo (N=135) | Olanzapine (N=131) | Open-label Risperidone LAI (N=560)
Acute stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 2 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Bipolar I disorder (Psychiatric disorders) | 2 | 5 | 1 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 4 | 1 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Female sterilisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 1
Hypomania (Psychiatric disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 6 | 17 | 6 | 16
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 0 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 3
Suicide attempt (Psychiatric disorders) | 2 | 2 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone LAI (N=132) | Placebo (N=135) | Olanzapine (N=131) | Open-label Risperidone LAI (N=560)
Agitation (Psychiatric disorders) | 3 | 6 | 6 | 25
Akathisia (Nervous system disorders) | 5 | 1 | 6 | 38
Amenorrhoea (Reproductive system and breast disorders) | 11 | 3 | 3 | 14
Anxiety (Psychiatric disorders) | 7 | 7 | 6 | 26
Fatigue (General disorders) | 5 | 0 | 11 | 10
Galactorrhoea (Reproductive system and breast disorders) | 7 | 0 | 0 | 13
Headache (Nervous system disorders) | 2 | 10 | 12 | 34
Hypersomnia (Nervous system disorders) | 2 | 4 | 10 | 4
Increased appetite (Metabolism and nutrition disorders) | 3 | 2 | 8 | 9
Influenza (Infections and infestations) | 1 | 9 | 1 | 7
Insomnia (Psychiatric disorders) | 21 | 24 | 13 | 87
Nausea (Gastrointestinal disorders) | 1 | 6 | 2 | 5
Somnolence (Nervous system disorders) | 8 | 4 | 16 | 16
Tremor (Nervous system disorders) | 5 | 6 | 5 | 28
Weight increased (Investigations) | 32 | 12 | 35 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days